CLINICAL TRIAL: NCT01704079
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Efficacy and Safety of CTAP101 Capsules to Treat Secondary Hyperparathyroidism in Subjects With Stage 3 or 4 Chronic Kidney Disease and Vitamin D Insufficiency
Brief Title: Safety and Efficacy of CTAP101 to Treat Secondary Hyperparathyroidism in Stage 3 or 4 CKD and Vitamin D Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OPKO IP Holdings II, Inc. (Industry)
Responsible Party: Sponsor
Organization: OPKO Health, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTAP101-CL-3002
Record Dates: First submitted 2012-10-06; First posted 2012-10-11 (Estimated); Results first posted 2016-08-17 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease; Hyperparathyroidism, Secondary; Vitamin D Deficiency
Keywords: Parathyroid Diseases; Renal Insufficiency; Kidney Failure, Chronic; Hyperparathyroidism, Secondary; Vitamin D; Hyperparathyroidism; Kidney Diseases; Kidney Failure; Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary; Vitamin D Deficiency; Parathyroid Diseases; Renal Insufficiency; Kidney Failure, Chronic; Hyperparathyroidism; Kidney Diseases | interventions — Calcifediol; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CTAP101 30 μg capsules (Active Comparator): 1 CTAP101 30 μg capsule daily at bedtime for 12 weeks, with a possible increase to 2 CTAP101 30 μg capsules daily at bedtime for study duration, if needed (26 weeks total). Subjects not requiring a dose increase after 12 weeks would receive 1 CTAP101 30 μg capsule and one sugar pill (to CTAP101 30 μg capsule) for weeks 13-26.
  Interventions: Drug: CTAP101 30 μg capsules; Other: Sugar pill to CTAP101 30 μg capsules
- Sugar pill to CTAP101 30 μg (Placebo Comparator): 1 sugar pill to CTAP101 30 μg capsule daily at bedtime for 12 weeks, with an increase to 2 sugar pills to CTAP101 30 μg capsules daily at bedtime for weeks 13-26.
  Interventions: Other: Sugar pill to CTAP101 30 μg capsules

INTERVENTIONS:
Drug: CTAP101 30 μg capsules — CTAP101 30 μg capsule taken daily at bedtime
  Other Names: Calcifediol
  Arms: CTAP101 30 μg capsules
Other: Sugar pill to CTAP101 30 μg capsules — Sugar pill capsule (placebo to CTAP101 30 μg capsule) taken daily at bedtime.
  Other Names: Placebo

SUMMARY:
This study will evaluate the efficacy of CTAP101 Capsules versus placebo in reducing intact parathyroid hormone (iPTH) by at least 30% from pretreatment baseline; safety and tolerability of CTAP101 will also be evaluated

DETAILED DESCRIPTION:
This is a phase 3, multi-center, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of CTAP101 Capsules administered for 26 weeks to treat SHPT in subjects ≥18 years of age with stage 3 or 4 CKD and vitamin D insufficiency. The study will be conducted at approximately 40 sites within the United States (US). Approximately 550 subjects will be screened to randomize approximately 210 eligible subjects, stratified by CKD stage (approximately 105 subjects in each stage) in a 2:1 ratio to receive either CTAP101 Capsules or matching placebo. An Interactive Voice Response System (IVRS) will provide study treatment group assignments using the computer-generated randomization code provided by the IVRS vendor. Subjects will receive an initial daily dose of 1 capsule (CTAP101 Capsules, 30 µg, or matching placebo) for the first 12 weeks. After l2 weeks (visit 8) and per pre-defined criteria, the dose may be increased in a blinded fashion by the IVRS with oversight by an independent medical monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Urinary albumin excretion ≤ 3000 mcg/mg of creatinine
2. Stage 3 or 4 CKD
3. Plasma iPTH: ≥ 85 pg/mL and < 500 pg/mL
4. Serum Ca: ≥ 8.4 mg/dL and < 9.8 mg/dL
5. Serum P: ≥ 2.0 mg/dL and < 5.0 mg/dL
6. Serum 25-hydroxyvitamin D: ≥ 10 ng/mL and < 30 ng/mL.
7. Stable dose of Vitamin D therapy ≤ 1600 IU/day and receiving same dose for at least 2 months

Exclusion Criteria:

1. History of kidney transplant or parathyroidectomy
2. Spot urine calcium:creatinine ratio > 0.2 (>200 mg/g Cr)
3. Current serious illness, such as malignancy, HIV, liver disease, cardiovascular event or hepatitis
4. Currently on dialysis
5. Use of pharmacological dose of ergocalciferol or cholecalciferol (≥ 50,000 IU mcg per month) during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Melnick, MD, Study Director — OPKO Renal
Locations (1):
- OPKO Renal, Bannockburn, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted at 45 investigational sites within the US. Subjects were enrolled and treated from 04 February 2013 through 13 August 2014.
Pre-assignment Details: Subjects were stratified by CKD stage and were randomized in a 2:1 ratio to receive a daily 30 μg oral dose of CTAP101 capsules (or matching placebo) for 12 weeks at bedtime. Subjects presenting on a regimen of bone metabolism therapy were to discontinue their prior treatment for at least 28 days' washout (except for bisphosphonates).
Period: Overall Study
Arm/Group | Sugar Pill to CTAP101 30 μg | CTAP101 30 μg Capsules
Started | 72 | 144
Entered Extension Study | 53 | 102
Completed | 58 | 121
Not Completed | 14 | 23
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Lost to Follow-up | 2 | 5
Not completed — Adverse Event | 4 | 7
Not completed — Protocol Violation | 1 | 0
Not completed — Subject noncompliance | 2 | 3
Not completed — Serum Calcium >/= 11.0 mg/dL, repeat con | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill to CTAP101 30 μg | CTAP101 30 μg Capsules | Total
Number analyzed (Participants) | 72 | 144 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (10.06) | 66.8 (10.90) | 66.3 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 71 | 110
  Male | 33 | 73 | 106
Region of Enrollment [Number; unit: participants]
  United States | 72 | 144 | 216

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in the Intent to Treat Population With Decrease in Plasma Intact Parathyroid Hormone (iPTH) of ≥30% From Pre-treatment Baseline
Description: Number of subjects in the intent to treat population attaining mean decrease in plasma intact Parathyroid Hormone (iPTH) of ≥30% from P\pre-treatment baseline in the efficacy assessment phase (EAP) referred to as responders
Time Frame: Approximately 6 months
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Sugar Pill to CTAP101 30 μg | CTAP101 30 μg Capsules
Number analyzed (Participants) | 72 | 144
participants | 5 | 49
Statistical Analysis 1: Comparison: Sugar Pill to CTAP101 30 μg vs CTAP101 30 μg Capsules; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Number of Participants in the Per Protocol Population With Decrease in Plasma Intact Parathyroid Hormone (iPTH) of ≥30% From Pre-treatment Baseline
Description: Number of subjects in the per protocol population attaining a mean decrease in plasma intact parathyroid hormone (iPTH) of ≥30% from pre-treatment baseline in the efficacy assessment phase (EAP), referred to as responders
Time Frame: Approximately 6 months
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Sugar Pill to CTAP101 30 μg | CTAP101 30 μg Capsules
Number analyzed (Participants) | 60 | 119
participants | 5 | 47
Statistical Analysis 1: Comparison: Sugar Pill to CTAP101 30 μg; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Subjects in the Intent to Treat Population With Normal Serum Total 25-hydroxyvitamin D
Description: Subjects in the intent to treat population with normal serum total 25-hydroxyvitamin D (>/= 30 ng/dL)
Time Frame: Approximately 6 months
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Sugar Pill to CTAP101 30 μg | CTAP101 30 μg Capsules
Number analyzed (Participants) | 72 | 144
participants | 5 | 120
Statistical Analysis 1: Comparison: Sugar Pill to CTAP101 30 μg vs CTAP101 30 μg Capsules; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Subjects in the Per Protocol Population With Normal Serum Total 25-hydroxyvitamin D
Description: Subjects in the per protocol population with normal serum total 25-hydroxyvitamin D (>/= 30 ng/mL)
Time Frame: Approximately 6 months
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Sugar Pill to CTAP101 30 μg | CTAP101 30 μg Capsules
Number analyzed (Participants) | 60 | 119
participants | 5 | 116
Statistical Analysis 1: Comparison: Sugar Pill to CTAP101 30 μg vs CTAP101 30 μg Capsules; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 6 months from randomization to end of therapy
Arm/Group | Sugar Pill to CTAP101 30 μg | CTAP101 30 μg Capsules
Serious Adverse Events (participants affected / at risk) | 11/72 | 22/144
Other Adverse Events (participants affected / at risk) | 18/72 | 32/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill to CTAP101 30 μg (N=72) | CTAP101 30 μg Capsules (N=144)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 3 (3)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Device malfunction (General disorders) | 0 (0) | 1 (1)
Cholelitiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Localized infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Myasthenia gravis crisis (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill to CTAP101 30 μg (N=72) | CTAP101 30 μg Capsules (N=144)
Constipation (Gastrointestinal disorders) | 4 (4) | 5 (5)
Oedema peripheral (General disorders) | 3 (3) | 9 (9)
Nasopharyngitis (Infections and infestations) | 1 (1) | 8 (8)
Gout (Metabolism and nutrition disorders) | 5 (5) | 6 (6)
Metabolic acidosis (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Hypertension (Vascular disorders) | 6 (6) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less